CLINICAL TRIAL: NCT00000733
Title: Phase I Pharmacokinetic and Tolerance Study of Ribavirin in Human Immunodeficiency Virus (HIV) - Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 035; 11011 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Ribavirin; T-Lymphocytes; Infusions, Intravenous; Immunologic Surveillance; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
To determine how fast ribavirin reaches the bloodstream, what concentration of ribavirin is reached in blood and how long it remains in the blood (pharmacokinetics) when given by different routes of administration. To find the maximum tolerated dose (MTD) of ribavirin. The effects of ribavirin on the immune system, and on the virus will be measured by T4 cell count and p24 antigen levels.

Early studies with ribavirin in patients with AIDS and AIDS related complex (ARC) have shown that ribavirin appears to inhibit the spread of the virus. Determination of how much and how often to give the drug will require further knowledge of the pharmacokinetics and toxicity of the drug in patients with AIDS or ARC and in chronic virus carriers who do not have symptoms.

DETAILED DESCRIPTION:
Early studies with ribavirin in patients with AIDS and AIDS related complex (ARC) have shown that ribavirin appears to inhibit the spread of the virus. Determination of how much and how often to give the drug will require further knowledge of the pharmacokinetics and toxicity of the drug in patients with AIDS or ARC and in chronic virus carriers who do not have symptoms.

Ribavirin is given to HIV-infected patients intravenously as a timed 30-min infusion at 1 of 5 single doses; 2 weeks later, the same doses are given orally in a single dose. Following at least 2 additional weeks, 6 patients are then given ribavirin at the lowest dose twice a day for 16 weeks. They are evaluated for tolerance and the next group is given a higher dose. Each successive group begins at 3-week intervals to receive doses that increase each day until the MTD is reached. Blood samples taken periodically during the treatment period and for 8 weeks after treatment is stopped are used to measure blood levels of ribavirin and to determine the effects of ribavirin on the HIV and immune system of the patients.

ELIGIBILITY:
Inclusion Criteria

Patients must be asymptomatic according to the following criteria:

* Normal neurologic exam.
* No unintentional weight loss of greater than 10 lbs. or more than 10 percent of usual body weight within 2 years prior to entering the study.
* No unexplained temperature above 38 degrees C on more than 5 consecutive days or on more than 10 days in any 30 days in the 2 years prior to expected entry into the study.
* No unexplained diarrhea defined by equal to or more than 3 liquid stools per day persisting more than 7 days within 2 years prior to expected entry into the study.
* No active hepatitis of any form. In addition, patients must not have previously had AIDS or an AIDS related illness.

Exclusion Criteria

Co-existing Condition:

Excluded:

* Temperature of greater than 37.8 degrees C.
* Development of an AIDS-defining opportunistic infection.
* Unexplained diarrhea defined by equal to or more than 3 liquid stools per day.
* Active hepatitis of any form.

Patients who have had oral candida infection documented by morphology, or by response to antifungal therapy, or oral hairy leukoplakia, or herpes zoster infection within 2 years of anticipated study entry at any time will be excluded. Patients with a prior history of a malignancy other than cutaneous basal cell carcinomas or cervical carcinoma in situ and patients with a significant chronic underlying medical illness that would impair continuous participation in the study will be excluded.

Prior Medication:

Excluded within 90 days of study entry:

* Immunomodulators.

Active alcohol or drug abuse sufficient in the investigator's opinion to prevent adequate compliance with the study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Study Completion 1991-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JJ Lertora, Study Chair
Locations (2):
- United States (2):
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana

REFERENCES:
- [Background] Lertora JJ, Rege AB, Lacour JT, Ferencz N, George WJ, VanDyke RB, Agrawal KC, Hyslop NE Jr. Pharmacokinetics and long-term tolerance to ribavirin in asymptomatic patients infected with human immunodeficiency virus. Clin Pharmacol Ther. 1991 Oct;50(4):442-9. doi: 10.1038/clpt.1991.162. PMID 1680594